CLINICAL TRIAL: NCT00000284
Title: Role of Metabolites in Nicotine Dependence (1)
Brief Title: Role of Metabolites in Nicotine Dependence (1) - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Minnesota (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09259-1; P50-09259-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Tobacco Use Disorder
Keywords: nicotine dependence
MeSH Terms: conditions — Tobacco Use Disorder

INTERVENTIONS:
Drug: Cotinine fumarate

SUMMARY:
The purpose of this study is to determine the effects of cotinine with or without a transdermal nicotine replacement on tobacco withdrawal symptoms.

DETAILED DESCRIPTION:
The purpose of this study was to determine the effects of a metabolite of nicotine, cotinine, on tobacco withdrawal symptoms. Cotinine has been shown to have psychoactive effects that are similar as well as different from those of nicotine, however, little research has been conducted examining the role cotinine plays in nicotine addiction. This study compared the effects of cotinine with the nicotine patch, and a combination thereof on tobacco withdrawal symptoms. The results showed that cotinine antagonizes the beneficial effects of the nicotine patch in reducing withdrawal symptoms.

ELIGIBILITY:
Inclusion Criteria:

Male or female subjects, aged 21-45 yrs inclusive, with a smoking history of at least 1 pack of cigarettes daily for at least 1 year. Subject must be in good health as verified by medical history, screening exam, and screening laboratory tests. Subject must provide written informed consent to participate in the study and be motivated to stop smoking for a short term.

Exclusion Criteria:

History of myocardial infarction, angina pectoris, sustained or episodic cardiac arrhythmias, symptomatic peripheral vascular disease, peptic ulcer disease or any other medical condition which the physician or investigator deems inappropriate for participation, insulin-dependent diabetes; pregnant or lactating or not using adequate birth control methods; requirement of any form of regular psychotropic medication (antidepressants, antipsychotics, or anxiolytics) and recent psychiatric history; chronic use of systemic steroids or antihistamines; skin sensitivity which would preclude use of a transdermal system; abuse of alcohol or any other recreational or prescription drug; use of any other tobacco products, including smokeless tobacco and nicotine products; previous use of transdermal nicotine system; inability to fulfill all scheduled visits and examination procedures throughout the study period.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1995-02; Study Completion 2001-12

PRIMARY OUTCOMES:
Subjective effects
Physiological effects
Performance effects

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] presented at Society of Research on nicotine and tobacco Psychopharmacology 1998. Presented at Society of Research on Nicotine and Tobacco Psychopharmacology (in press)
- [Derived] Campos CM, Mehran R, Capodanno D, Owen R, Windecker S, Varenne O, Stone GW, Valgimigli M, Hajjar LA, Kalil Filho R, Oldroyd K, Morice MC, Urban P, Abizaid A. Risk Burden of Cancer in Patients Treated With Abbreviated Dual Antiplatelet Therapy After PCI: Analysis of Multicenter Controlled High-Bleeding Risk Trials. Circ Cardiovasc Interv. 2024 Apr;17(4):e013000. doi: 10.1161/CIRCINTERVENTIONS.122.013000. Epub 2024 Apr 16. PMID 38626080